CLINICAL TRIAL: NCT05114837
Title: Phase I/II First-in-Human Trial With CAR19 Regulatory T Cells (CAR19-tTreg) in Adults With Relapsed/Refractory CD19+ B Acute Lymphocytic Leukemia
Brief Title: Ph I/II Study of CAR19 Regulatory T Cells (CAR19-tTreg) for R/R CD19+ B-ALL
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: replaced with a new IND and protocol
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021LS012; MT2021-02 (Other: University of Minnesota)
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma Leukemia
Keywords: CAR19-tTreg
MeSH Terms: interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Evaluate the safety profile and potential efficacy of allogeneic CAR19 regulatory T cells (CAR19-tTreg)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I/II (Experimental): Determine the maximum tolerated dose (MTD) of CAR19-tTreg. It will be administered in a single dose after high dose lymphodepleting chemotherapy to promote adoptive transfer. First dose of 1.0 x 10 6 CAR19-tTreg/kg recipient body weight (dose level 1).The subsequent doses are 3.0, 10.0 and 30.0 x 10 6 CAR19- tTreg/kg. PHASE II Expand trial on maximum tolerated dose (MTD) of CAR19-tTreg from Phase I. It will be administered in a single dose after high dose lymphodepleting chemotherapy to promote adoptive transfer.The CAR19-tTreg/kg dose is to be determined.
  Interventions: Drug: allogeneic CAR19 regulatory T cells (CAR19-tTreg); Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: allogeneic CAR19 regulatory T cells (CAR19-tTreg) — A single dose administration of CAR19-tTreg
Drug: Fludarabine — Fludarabine 30 mg/m^2 is administered as an intravenous (IV) infusion per institutional guidelines once a day on 4 consecutive days (Day -5, Day -4, Day -3 and Day -2)
  Other Names: FLUDARA
Drug: Cyclophosphamide — Cyclophosphamide 500 mg/m^2 is administered as an IV infusion per institutional guidelines once a day on 2 consecutive days (Day -5, and Day -4)
  Other Names: CYTOXAN

SUMMARY:
This is a single-center, single-arm, interventional phase I/II trial to evaluate the safety profile and potential efficacy of allogeneic CAR19 regulatory T cells (CAR19-tTreg) in adults with relapsed/refractory (R/R) CD19+ B Acute Lymphocytic Leukemia (B-ALL).

The study consists of two components. The dose finding component is a modified version of a Phase I trial and the extended component is a modified Phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of R/R CD19+ B-ALL after failure of standard of care therapies with CD19 expression on blasts confirmed by flow cytometry or immunohistochemistry and meeting one or more of the following criteria:

  1. Primary induction failure with no complete remission after ≥2 cycles of induction chemotherapy/immunotherapy, or
  2. First relapse with no CR after 1 cycle of induction therapy, or
  3. Second or greater relapse, or
  4. Ph+ ALL and failure or intolerance to three lines of tyrosine kinase inhibitors (TKI) assuming one or more of the above criteria are also met.
* Karnofsky performance status (KPS) ≥70% at screening
* Adequate organ function is defined as:

  1. Renal: Calculated estimated glomerular filtration rate greater than or equal to50 mL/min/1.73 m2
  2. Hepatic: ALT and AST less than 3x upper limit of normal (ULN), and bilirubin less than2x ULN (exception, patients with Gilbert syndrome, total less than 3 x ULN and direct less than 1.5 x ULN)
  3. Cardiac: Left ventricular ejection fraction (LVEF) greater than 45% by echocardiogram
  4. Pulmonary: SpO2 greater than 92% on room air
* Use of antiproliferative chemotherapy more than 2 weeks prior to enrollment and blinatumomab more than 4 weeks prior to enrollment
* Patients with relapsed disease after prior allogeneic transplantation may be considered. In addition to the eligibility criteria otherwise listed, this subgroup must be more than 3 months from allogeneic hematopoietic stem cell transplant (HSCT), off immune suppressive therapy (e.g., calcineurin inhibitor, glucocorticoid, sirolimus) at least 4 weeks without GVHD.
* Patients who received prior CAR-T therapy are eligible if more than 2 months after CAR-T infusion and CD19 expression is confirmed at the most recent relapse and all other criteria are met
* Voluntary informed consent by the patient for treatment and follow-up for 15 years after treatment.

Exclusion Criteria:

* Availability of a FDA approved CAR T cell therapeutic targeting CD19+ B-ALL (patients eligible for but unable to receive FDA approved CAR T cells based on insurance limitations, may be eligible for the proposed trial)
* Use of pharmacological immunosuppressive agents within 2 weeks (with the exception of physiologic or stress dose glucocorticoid replacement) or anti-T cell antibodies within 2 months of study participation
* Diagnosis of Burkitt lymphoma
* Diagnosis of active central nervous system (CNS) leukemia
* Known allergy to manufacturing components: human albumin or dimethylsulfoxide (DMSO)
* History of HIV infection on anti-retroviral therapy
* Positive for hepatitis B or hepatitis C
* Active uncontrolled bacterial, fungal, or viral infections - all prior infections must have resolved or be improving following optimal therapy
* Active autoimmune disease requiring immunosuppressive therapy
* Class II or greater New York Heart Association Functional Classification criteria or serious cardiac arrhythmias likely to increase the risk of cardiac complications of cytokine therapy (e.g. ventricular tachycardia, or supraventricular tachyarrhythmia requiring chronic therapy)
* Females who are pregnant or breastfeeding
* Unstable angina, arrhythmias, evidence of acute ischemia or conduction system abnormalities by electrocardiogram (ECG) or myocardial infarction in prior to 2 months
* Use of other investigational agents within 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Dose Finding of CAR19-tTregs | 28 days after CAR19-tTregs administrations
  To identify the MTD of CAR19-tTregs defined asthe dose level that most closely corresponds to a dose limiting toxicity rate(DLT) less than or equal to 25%. Using grade 3-5 Common Terminology Criteria for Adverse Events version 5 (CTCAEv5) Statistical Analysis: The proportion of patients with ORR, CR and adverse events by day 28 will be estimated by simple proportions with 95% confidence intervals
Measure CAR19-tTregs efficacy | 28 days after CAR19-tTregs administrations
  Efficacy estimate as measured by overall response rate

SECONDARY OUTCOMES:
Incidence of CR | 28 days after CAR19-tTregs administrations
  Report number patients that achieved complete response (CR)
Incidence of grade 3-4 cytokine release syndrome (CRS) | 28 days after CAR19-tTregs administrations
  Evaluated using the American Society of Transplantation and Cellular Therapy (ASTCT) CRS consensus grading system
Incidence of immune cell associated neurotoxicity syndrome (ICANS) | 28 days after CAR19-tTregs administrations
  Report the count of neurotoxicities based on the ICANS system.
Incidence of relapse in patients achieving complete response (CR) | 1 year after treatment
  Report the count of relapses out of those that achieved complete reponse
Incidence of relapse in patients achieving complete (CR) | Day +100 after treatment
  Report the count (as proportions) of relapses out of those that achieved complete re
Probability of survival and event free survival | 6 months
  The analysis of overall survival will use death as the event, and the analysis of event-free survival will use the earliest of no response, relapse, or death as the event. Patients who do not have an event will have their data censored for the analyses at the date at which they were last known to be alive. Finally, probabilities will be measured using Kaplan-Meier curves
Probability of survival and event free survival | 1 year
  The analysis of overall survival will use death as the event, and the analysis of event-free survival will use the earliest of no response, relapse, or death as the event. Patients who do not have an event will have their data censored for the analyses at the date at which they were last known to be alive. Finally, probabilities will be measured using Kaplan-Meier curves

CONTACTS AND LOCATIONS:
Overall Officials: Bachanova Veronika, MD, Principal Investigator — Masonic Cancer Center, Univeristy of Minnesota
Locations (1):
- Masonic Cancer Center - University of Minnesota, Minneapolis, Minnesota, United States